CLINICAL TRIAL: NCT00352560
Title: Electrophysiological Effects of Irbesartan in Patients With Paroxysmal Atrial Fibrillation (AF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV131-235
Record Dates: First submitted 2006-07-12; First posted 2006-07-14 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2008-06

CONDITIONS: Atrial Fibrillation
Keywords: Patients with Paroxysmal Atrial Fibrillation (PAF)
MeSH Terms: conditions — Atrial Fibrillation | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Irbesartan
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Irbesartan — Tablets, Oral, 300 mg, once daily, 30 days.
  Other Names: Avapro
  Arms: A
Drug: Placebo — Tablets, Oral, 0 mg, once daily, 30 days.
  Arms: B

SUMMARY:
The main purpose of the study is to compare the mean AERP between treatment groups based on the hypothesis that in subjects with paroxysmal AF, Irbesartan prevents electrophysiological remodeling resulting in a prolonged atrial effective refractory period relative (AERP) to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent PAF with indication for catheter ablation

Exclusion Criteria:

* Struct. Cardiopathy
* Mitral valve disease
* VEF<40%
* Myocardiopathy
* LVH
* cardiac surgery
* AF reversible
* QT c>450
* Recent MI/stroke, severe HTN
* Requirement of ACEI/ARBs
* Coronary synd., HTA, liver disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2006-07; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Irbesartan effect on duration of Atrial Effective Refractory Period (AERP) in paroxysmal AF (PAF) patients. | The measures are taken after 31 days of irbesartan treatment

SECONDARY OUTCOMES:
Irbesartan effect on A Function RP | The measures are taken after 31 days of irbesartan treatment
Irbesartan effect on atrial conduction intervals after basal & extra-stimuli, in PAF patients | The measures are taken after 31 days of irbesartan treatment
Refractoriness dispersion | The measures are taken after 31 days of irbesartan treatment

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Sanchez Zamorano, MD, Study Director — Medical Department, Bristol-Myers Squibb
Locations (1):
- Local Institution, Madrid, Spain